CLINICAL TRIAL: NCT02992457
Title: Study of the Safety and Efficacy of Sofosbuvir-Based Regimens in the Treatment of Egyptian Patients With and Without Post-hepatitis C Cirrhosis
Brief Title: Safety and Efficacy of Sofosbuvir-Based Regimens in the Treatment of Egyptian Patients With Hepatitis C Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Asem Elfert
Record Dates: First submitted 2016-12-06; First posted 2016-12-14 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; Ribavirin; peginterferon alfa-2a; Simeprevir; daclatasvir; paritaprevir; ledipasvir, sofosbuvir drug combination; Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Sof-Riba (Active Comparator): Sofosbuvir ribavirin 6 months.
  Interventions: Drug: Sofosbuvir; Drug: Ribavirin
- Sof- Riba- Pegylated interferon (Active Comparator): Sofosbuvir, Ribavirin and Pegylated-interferon alfa-2a 3 months
  Interventions: Drug: Sofosbuvir; Drug: Ribavirin; Drug: Pegylated-interferon alfa-2a
- Sof- Olysio (Active Comparator): Sofosbuvir and simeprevir for 3 months.
  Interventions: Drug: Sofosbuvir; Drug: Simeprevir
- Sof- Dacla (Active Comparator): Sofosbuvir and Daclatasvir for 3 months.
  Interventions: Drug: Sofosbuvir; Drug: Daclatasvir
- Harvony (Active Comparator): Sofosbuvir and ledipasvir for 3 months
  Interventions: Drug: Sofosbuvir and Ledipasvir
- Ritaprevir, paritaprevir, ombetasvir (Active Comparator): Querevo for 3 months
  Interventions: Drug: Ritaprevir, paritaprevir, ombetasvir
- Salvage therapy (Active Comparator): sofosbuvir, daclatasvir, simeprevir,ribavirin or sofosbuvir and querevo
  Interventions: Drug: Salvage therapy

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 mg daily.
  Other Names: sovaldi , mpiviropack
  Arms: Sof- Dacla; Sof- Olysio; Sof- Riba- Pegylated interferon; Sof-Riba
Drug: Ribavirin — Ribavirin 1000-1200 mg daily
  Other Names: Rebetol, Riba
  Arms: Sof- Riba- Pegylated interferon; Sof-Riba
Drug: Pegylated-interferon alfa-2a — Pegylated interferon alfa-2a once weekly for 3 months
  Other Names: peginteron, pegasys
  Arms: Sof- Riba- Pegylated interferon
Drug: Simeprevir — Olysio once daily.
  Other Names: Olysio
  Arms: Sof- Olysio
Drug: Daclatasvir — Dakla once daily for three months.
  Other Names: Daklatasvir, Dakla
  Arms: Sof- Dacla
Drug: Ritaprevir, paritaprevir, ombetasvir — Querevo for three months
  Other Names: querevo
  Arms: Ritaprevir, paritaprevir, ombetasvir
Drug: Sofosbuvir and Ledipasvir — Once daily for three months
  Other Names: Harvony
  Arms: Harvony
Drug: Salvage therapy — three months in repeated treatment failure
  Other Names: Sofosbuvir,simeprevir, daclatasvir, ribavirin or sofosbuvir and querevo
  Arms: Salvage therapy

SUMMARY:
Egypt has the highest prevalence of hepatitis C virus (HCV) in the world, estimated nationally at 14.7%. Genotype 4 (and subtype 4a in particular) dominates the HCV epidemic in Egypt. For decades the antiviral therapy of chronic HCV infection was based on the administration of Interferon(IFN), initially alone and then in combination with Ribavirin (RBV), but this regimen was effective in only 50% of patients with genotype 1, with significant side effects.

DETAILED DESCRIPTION:
Egypt has the highest prevalence of hepatitis C virus (HCV) in the world, estimated nationally at 14.7%. Genotype 4 (and subtype 4a in particular) dominates the HCV epidemic in Egypt. For decades the antiviral therapy of chronic HCV infection was based on the administration ofInterferon(IFN), initially alone and then in combination with Ribavirin (RBV), but this regimen was effective in only 50% of patients with genotype 1, with significant side effects. The introduction of direct acting antiviral agents, in particular sofosbuvir (SOF), has revolutionized the treatment for chronic hepatitis C virus.

ELIGIBILITY:
Inclusion Criteria:

* • HCV infection

  * Adult patients, 18years and older.

Exclusion Criteria:

* • Child score > 12

  * Severe Renal impairment
  * Pregnant and lactating women
  * HCC or other malignant neoplasms
  * Co-infection with human immunodeficiency virus (HIV)
  * Co-infection with hepatitis B virus (HBV)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with sustained virological response. | 2 months
  The number of patients achieving SVR

CONTACTS AND LOCATIONS:
Overall Officials: Asem Elfert, Prof, Study Chair — Tanta university hospital; Lobna Abo ALi, Ass Prof, Study Chair — Tanta university hospital; Sabry Abou Saif, Ass Prof, Study Chair — Tanta university hospital; Taher Eldemerdash, Prof, Study Chair — Tanta University hospital; Hala M Elsabagh, Prof, Study Chair — Tanta University hospital; Mohamed Elkassas, Lecturer, Study Chair — Helwan University; Eslam Esmail, Ass Lecturer, Study Chair — Tanta University; Sherief Abd-Elsalam, Principal Investigator — Tanta University
Locations (2):
- Egypt (2):
  - Sherief Abd-Elsalam, Tanta
  - Tanta university hospital, Tanta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Said EM, Abdulaziz BA, El Kassas M, El Attar IH, Emadeldeen M, Abd-Elsalam SM. High success rates for the use of sofosbuvir/ombitasvir/paritaprevir/ritonavir + ribavirin and sofosbuvir/simeprevir/daclatasvir + ribavirin in retreatment of chronic hepatitis C infection after unsuccessful sofosbuvir/daclatasvir therapy: a real-life experience. Arch Virol. 2020 Jul;165(7):1633-1639. doi: 10.1007/s00705-020-04639-x. Epub 2020 Apr 30. PMID 32356185
- [Derived] Ahmed OA, Kaisar HH, Badawi R, Hawash N, Samir H, Shabana SS, Fouad MHA, Rizk FH, Khodeir SA, Abd-Elsalam S. Efficacy and safety of sofosbuvir-ledipasvir for treatment of a cohort of Egyptian patients with chronic hepatitis C genotype 4 infection. Infect Drug Resist. 2018 Mar 1;11:295-298. doi: 10.2147/IDR.S153060. eCollection 2018. PMID 29535545